CLINICAL TRIAL: NCT00112021
Title: A Phase 2B, Randomized, Double-Blinded, Placebo-Controlled, Dose Ranging, Multicenter Study to Examine the Effect of Pramlintide on Body Weight and Its Safety and Tolerability in Obese Subjects
Brief Title: A Study to Examine the Effect of Pramlintide on Body Weight and Its Safety and Tolerability in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 137OB-201
Record Dates: First submitted 2005-05-27; First posted 2005-05-30 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: obesity; weight loss; Amylin; pramlintide; Symlin
MeSH Terms: conditions — Obesity; Weight Loss | interventions — pramlintide

ARMS (2):
- Pramlintide Acetate (Experimental)
  Interventions: Drug: pramlintide acetate
- Placebo (Placebo Comparator)

INTERVENTIONS:
Drug: pramlintide acetate
  Other Names: Pramlintide acetate injection (Pramlintide (0.6 mg/mL)) is a clear, colorless, sterile solution for SC injection
  Arms: Pramlintide Acetate

SUMMARY:
This is a study to examine the effect of pramlintide on body weight and its safety and tolerability in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Is obese with a body mass index (BMI) >=30 kg/m^2 to <=50 kg/m^2, and has been obese for at least one year before screening.
* Usually consumes at least three major meals (morning, midday, and evening) each day.

Exclusion Criteria:

* Is currently enrolled in a formal weight-loss program.
* Has had liposuction within 1 year before screening or is planning to have liposuction during the study.
* Has received any investigational drug within 3 months before screening.
* Has previously participated in a study using pramlintide.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2005-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To examine the effect of pramlintide on body weight in obese subjects | Approximately 16 weeks
To examine the safety and tolerability of pramlintide in obese subjects | Approximately 16 weeks

SECONDARY OUTCOMES:
To investigate the effect of pramlintide in obese subjects on anthropometric and fasting/postprandial humoral metabolic parameters | Approximately 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (21):
- United States (21):
  - Research Site, Chula Vista, California
  - Research Site, San Diego, California
  - Research Site, Walnut Creek, California
  - Research Site, Miami, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Edina, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Olympia, Washington

REFERENCES:
- [Derived] Smith SR, Aronne LJ, Burns CM, Kesty NC, Halseth AE, Weyer C. Sustained weight loss following 12-month pramlintide treatment as an adjunct to lifestyle intervention in obesity. Diabetes Care. 2008 Sep;31(9):1816-23. doi: 10.2337/dc08-0029. Epub 2008 Jun 20. PMID 18753666